CLINICAL TRIAL: NCT01474824
Title: Validation of the Nexfin Non-invasive Cardiac Output Monitor in Patients Undergoing Hip Fracture Repair
Brief Title: Validation of Nexfin Cardiac Output in Elderly Patients With Hip Fracture
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit sufficient participants
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 11090; 11/SW/0288 (Other: NRES)
Record Dates: First submitted 2011-10-14; First posted 2011-11-18 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Hip Fractures; Anesthesia
Keywords: Cardiac output; Stroke volume
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Measurement of how much blood the heart pumps may be useful in guiding how much intravenous fluid to give patients during surgery. The current monitors either require special drips (arterial and/or central lines) or a probe inserted into the oesophagus (food pipe) which may limit their use. Newer monitors are available which are completely non-invasive and seem to work well in younger patients. Patients with hip fracture are elderly and frail. The investigators wish to see whether the newer non-invasive monitor works well enough compared to the current monitors in this group of patients. If it does this may allow more of these patients to be monitored in this way.

DETAILED DESCRIPTION:
The investigators wish to compare the accuracy of the newer, non-invasive monitor (Nexfin) against a more established minimally invasive monitor (LiDCO). The LiDCO has a calibration system which allows the absolute accuracy of the Nexfin to be established.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 80
* Able to give their own informed consent

Exclusion Criteria:

* Severe valvular heart disease
* Taking lithium

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing surgical repair of hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Bias and limits of agreement of Nexfin recorded cardiac output compared with LiDCOplus | During anaesthesia period of surgery - measurements will be complete within 30 minutes of starting anaesthesia
  Analysis of agreement between Nexfin cardiac output and the calibrated cardiac output measured by LiDCOplus

SECONDARY OUTCOMES:
Bias and limits of agreement for change in cardiac output measured by Nexfin compared with LiDCO | During anaesthesia period of surgery - measurements will be complete within 30 minutes of starting anaesthesia
  Comparison of relative changes in cardiac output recorded by Nexfin and LiDCO in response to intra-anaesthesia / intra-operative events (fluid administration, drug administration)
Utility of Nexfin monitor | Intra-operative - average duration about 1 hour
  Proportion of time during anaesthesia and surgery when a valid signal is obtained from the Nexfin device.
Adverse events associated with Nexfin monitor | Intra-operative - average duration about one hour
  Recording of adverse events associated with use of the Nexfin monitor

CONTACTS AND LOCATIONS:
Overall Officials: Iain K Moppett, DM FRCA MRCP, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals, Nottingham, Notts
  - Brighton and Sussex University Hospitals, Brighton, Sussex

REFERENCES:
- [Background] Wiles MD, Whiteley WJ, Moran CG, Moppett IK. The use of LiDCO based fluid management in patients undergoing hip fracture surgery under spinal anaesthesia: neck of femur optimisation therapy - targeted stroke volume (NOTTS): study protocol for a randomized controlled trial. Trials. 2011 Sep 28;12:213. doi: 10.1186/1745-6215-12-213. PMID 21955538